CLINICAL TRIAL: NCT06670092
Title: Effect of Vojta Therapy on Motor Control in Children With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, Principal investigator, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09/2024
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention-Deficit/Hyperactivity Disorder; Vojta Therapy; balance; postural control; visual motor coordination; manipulative skills
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): This group is treated according to Vojta therapy
  Interventions: Other: Vojta Therapy
- Control group (Other): This group does not receive treatment
  Interventions: Other: No intervetion

INTERVENTIONS:
Other: Vojta Therapy — The intervention is carried out using Vojta therapy for one month, with one session per day, 5 days a week. This therapy is carried out by an expert physiotherapist. Vojta therapy is a non-experimental, painless, non-invasive therapy with no adverse effects, which is based on triggering repeated motor reactions or innate movement patterns (reflex locomotion patterns) in the trunk and limbs based on defined stimuli and starting from specific postures.
  Both groups will undertake a pre-treatment assessment, a post-treatment assessment at the end of the one-month intervention period, and a final follow-up assessment one month after the end of the intervention.
  Arms: Experimental group
Other: No intervetion — No intervetion group
  Other Names: No intervention group
  Arms: Control group

SUMMARY:
ADHD is generally associated with significant comorbidities including motor disorders in up to 96% of cases. Within these, disturbances of balance and motor coordination that interfere with school learning and daily activities are present in 47% of school children with ADHD. Therefore, the aim of this research is to determine whether Vojta therapy is beneficial for the improvement of balance, postural control, hand-eye coordination and manipulative motor skills in children with ADHD, hyperactive and/or combined, aged 6-12 years.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of Attention Deficit Hyperactivity Disorder (ADHD) of the combined or hyperkinetic type.
2. Be between 6 and 12 years of age.
3. Be under treatment with methylphenidate.
4. IQ of 100 or higher.
5. Have a normal neurological examination.
6. Not dysmorphic.
7. Not have received specific physiotherapy treatment for the improvement of balance and postural control in the two months prior to inclusion in the study.

Exclusion Criteria:

1. Present a diagnosis of ADHD comorbid with other neuropsychiatric pathologies.
2. Have a history of neurological or musculoskeletal disorders that are linked to a deficit in balance and/or postural control.
3. Be under treatment with atomoxetine.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Sensory organisation test (NEUROCOM dynamic posturology) | 15 minutes
  This test is a commonly used research tool in the assessment of the sensory organisation of postural control and has previously been used in children. The system's force platform provides data on the movement of the centre of gravity. Both the platform and the environment can move in response to the anteroposterior displacement of the child's body under certain conditions of sensory override or conflict. The child is asked to stand upright, barefoot, with arms alongside the body, feet placed in a certain position on the platform, for 20sec, trying to remain as stable as possible during the 3 trials of each of the 6 conditions of the SOT. For their safety, the child shall be restrained by a harness. In each test, the system compares the child's displacement with its theoretical limits of stability, generating a score. The higher the value, the better the stability. The software also calculates an overall score from the scores obtained in each of the 6 conditions

SECONDARY OUTCOMES:
Paediatric Balance Scale | 15 minutes
  This is a clinical scale used to assess balance in children aged 5 to 15 years. It consists of 14 items (each rated at 0-4 points), is easy to perform, does not require specialised equipment and takes less than 15 minutes to complete. It is considered the paediatric alternative to the Berg Balance Scale in school-aged children with mild to moderate motor impairment, with good intra- and inter-observer reliability.
Bruininks-Oseretsky Test (abbreviated version) | 10 minutes
  This test assesses agility and speed in running, balance, bilateral coordination, strength, coordination and response speed of the upper limb, visual-motor control and speed and dexterity of the upper limb. This test has been used in the ADHD population.
Paediatric Quality of Life Questionnaire | 10 minutes
  It is a widely studied and used instrument, designed for children, which has a generic module for paediatric quality of life, which also has specific modules for various chronic diseases and clinical situations. The different existing versions will be used depending on the age of the child (questionnaire for children aged 5 to 7 years and questionnaire for children aged 8 to 12 years) validated and translated into Spanish. Both questionnaires can be administered to the child or to the parents.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes